CLINICAL TRIAL: NCT02306603
Title: Outcomes of Endoscopic Resection of Mucosal and Submucosal Lesions in the Duodenum and Ampulla
Brief Title: Long-term Outcomes of Endoscopic Resection (ER) of Lesions of the Duodenum and Ampulla
Acronym: OERDA
Status: Recruiting | Type: Observational
Sponsor: Professor Michael Bourke (Other)
Responsible Party: Sponsor-Investigator, Professor Michael Bourke, Director of Gastrointestinal Endoscopy, Western Sydney Local Health District
Organization: Western Sydney Local Health District (Other)
Other Study IDs: HREC 2014/5/4.3 (3972)
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Adenoma, Villous
MeSH Terms: conditions — Adenoma, Villous | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Endoscopic Mucosal Resection: Patients who are referred for Endoscopic Mucosal Resection of Duodenal and Ampullary Lesions will be included in this cohort.
  Interventions: Procedure: Endoscopic Mucosal Resection

INTERVENTIONS:
Procedure: Endoscopic Mucosal Resection

SUMMARY:
This research project, 'Outcomes of endoscopic resection of mucosal and submucosal lesions in the duodenum and ampulla'. The research project is aiming to determine the most effective and safe way to remove such lesions.

DETAILED DESCRIPTION:
Endoscopic resection (ER) of superficial lesions of the duodenum and ampulla is a safe and effective surgery sparing modality in experienced hands. It is often curative of dysplastic lesions and is associated with minimal complications and high patient acceptance (1-5). Westmead Hospital has accumulated a significant amount of experience in the removal of such lesions; however, there is limited research to document the long term outcomes of patients undergoing endoscopic resection.The purpose of this study is to evaluate the long-term outcomes of ER of superficial lesions of the duodenum and ampulla.

ELIGIBILITY:
Inclusion Criteria:

* Duodenal and ampullary lesion > 10mm

* Lesion limited to the mucosal and/or submucosal layer (T1 lesion)
* Aged 18 years or older

Exclusion Criteria:

* Lesion less than 10mm
* Duodenal or ampullary lesion involves the muscularis propria (T2 lesion) on other staging modalities such as endoscopic ultrasonography (EUS)
* Aged younger than 18 years

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have Duodenal and ampullary adenomas which are amendable to Endoscopic Mucosal Resection
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-10; Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Observed procedural data: Number of Participants with Adverse Events as a Measure of Safety and Tolerability Outcomes | 14 days

SECONDARY OUTCOMES:
Analysis of the costs of this procedure compared to previous treatments | 14 days
  Perform cost-utility analyses comparing different treatment approaches for duodenal and ampullary lesions

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Bourke, MBBS, Principal Investigator — Western Sydney Local Health District
Locations (1):
- Westmead Hospital Endoscopy Unit, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Gupta S, Craciun A, Wang H, Whitfield A, Gauci J, O'Sullivan T, Cronin O, Abu Arisha M, Klein A, Lee EYT, Burgess NG, Bourke MJ. Hybrid resection versus conventional resection for laterally spreading lesions of the papilla. Gastrointest Endosc. 2024 Mar;99(3):428-436. doi: 10.1016/j.gie.2023.10.034. Epub 2023 Oct 17. PMID 37858758
- [Derived] Wang H, Sidhu M, Gupta S, Cronin O, O'Sullivan T, Whitfield A, Burgess NG, Bourke MJ. Cold snare EMR for the removal of large duodenal adenomas. Gastrointest Endosc. 2023 Jun;97(6):1100-1108. doi: 10.1016/j.gie.2023.01.040. Epub 2023 Jan 28. PMID 36720290
- [Derived] Sidhu M, Fritzsche JA, Klein A, Shahidi N, Vosko S, van Hattem WA, Tate DJ, Bourke MJ. Outcomes of thermal ablation of the defect margin after duodenal endoscopic mucosal resection (with videos). Gastrointest Endosc. 2021 Jun;93(6):1373-1380. doi: 10.1016/j.gie.2020.11.024. Epub 2020 Dec 4. PMID 33285144
- [Derived] Klein A, Qi Z, Bahin FF, Awadie H, Nayyar D, Ma M, Voermans RP, Williams SJ, Lee E, Bourke MJ. Outcomes after endoscopic resection of large laterally spreading lesions of the papilla and conventional ampullary adenomas are equivalent. Endoscopy. 2018 Oct;50(10):972-983. doi: 10.1055/a-0587-5228. Epub 2018 May 16. PMID 29768645